CLINICAL TRIAL: NCT05914142
Title: Study on the Safety and Effectiveness of Varian ProBeam Proton Therapy Equipment in the Treatment of Solid Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Concord Cancer Center (Other)
Collaborators: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Varian, a Siemens Healthineers Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSQX-2022-046-02
Record Dates: First submitted 2023-05-09; First posted 2023-06-22 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Solid Tumor; Radiation Therapy; Proton Therapy
Keywords: varian; Probeam
MeSH Terms: interventions — Proton Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Proton radiation therapy group (Experimental): Experimental: single-arm objective performance criteria, OPC
  Interventions: Device: Proton radiation therapy

INTERVENTIONS:
Device: Proton radiation therapy — Radiation: Proton Therapy System (ProBeam)

SUMMARY:
This study is a clinical trial of prospective, single-arm objective performance criteria. This trial will be conducted in clinical trial sites with a total of 47 subjects enrolled. All of subjects will be treated with radiation therapy using the medical device Varian ProBeam Proton Therapy System (ProBeam), aim to compare the data with objective performance criteria (OPC) to evaluate the effectiveness and safety of ProBeam radiotherapy system for oncology patients, providing a clinical basis for the medical device registration.

DETAILED DESCRIPTION:
Oncology patients, including tumors of the nervous system, head and neck, chest, abdomen, spine, pelvic cavity, limbs and other tumors. The screening period from informed consent to enrollment is expected to be 4 weeks, while the treatment period is 1 to 8 weeks. The period after the last treatment is divided into short-term follow-up and long-term follow-up, in which short-term follow-up will be 3 months after the end of the last treatment. Total expected participation for each subject from screening to the completion of short-term follow-up is a maximum duration of 12 weeks + 3 months. Long-term follow-up continues after the end of short-term follow-up until the 5th year after the end of the last radiotherapy session.

ELIGIBILITY:
Inclusion Criteria:

1.18≤ age≤ 80 years;

2.First-diagnosed patients with tumors of the nervous system, head and neck, chest, abdomen, spine, pelvic cavity, limbs, etc. by tissue/cell pathology;

3.ECOG physical condition is graded as 0 to 2;

4.Women of childbearing had negative results in the blood pregnancy test (Human Chorionic Gonadotropin, HCG) 7 days prior to the first treatment;

5.The subject or subject's guardian is able to understand the purpose of the study, demonstrate sufficient compliance with the protocol and sign informed consent form

Exclusion Criteria:

1. The subject with radiotherapy contraindications, including the known genetic tendencies that increase the sensitivity of normal tissue radiotherapy or the accompanying diseases that lead to hypersensitivity to radiotherapy;
2. The subject with other uncontrolled tumors except that to be treated according to medical history or the investigator's estimation, or with other malignant tumors within five years prior to enrollment;
3. Implanted pacemakers or other metal prosthesis within the scope of proton therapy;
4. Other situations that investigator determines not suitable for enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-07-04 (Actual); Study Completion 2023-07-04 (Actual)

PRIMARY OUTCOMES:
tumor disease control rate reaches the objective performance criteria | 3 months ± 7 days after the last treatment
  After treatment, CR, PR, SD is considered disease control; Percentage of subjects who developed disease control 3 months after the end of the last radiotherapy session.
CTCAE level 3 toxic reaction ratio is lower than the acceptable value | started from subject enrollment to 3 months ± 7 days after the last treatment, up to 5 months
  The proportion of subjects whose toxicity reaction is level 3 during the clinical trial period. The researchers record AE that appeared during the clinical trial cycle and grade it according to CTCAE 5.0
CTCAE level 4 and 5 toxic reaction ratio is acceptable value | the entire clinical trial ( until 3 months after last treatment)
  The proportion of subjects with toxic reactions of levels 4 and 5 during the clinical trial period.The researchers record AE that appeared during the clinical trial cycle and grade it according to CTCAE 5.0)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | screening, 1 months ± 7 days, 2 months ± 7 days, 3 months ± 7 days after the last treatment
  The appearance of CR or PR after treatment is considered objective response, Percentage of subjects who experienced objective response at each point in time after the end of the last treatment
Duration of Response (DOR) | screening, 1 months ± 7 days, 2 months ± 7 days, 3 months ± 7 days after the last treatment
  The duration of the tumor's first assessment as CR or PR, until the first assessment of PD or death due to any cause.
Disease Control Rate (DCR) | screening, 1 months ± 7 days, 2 months ± 7 days, 3 months ± 7 days after the last treatment
  CR, PR, SD for disease control after treatment
tumor markers (if applicable), Tumor-specific symptoms | screening, 1 months ± 7 days, 2 months ± 7 days, 3 months ± 7 days after the last treatment
  Tumor markers are examined and the researchers determine the clinical significance of reporting changes in tumor markers (before and after radiation therapy). The symptoms may be recorded according to the disease, and the researchers determine the clinical significance of reporting symptoms (before and after radiation therapy)
actual situation of Product usability evaluation (ProBeam system, Oncology Information system (OIS), Treatment plan system (Eclipse)) | screening, 1 months ± 7 days, 2 months ± 7 days, 3 months ± 7 days after the last treatment
  Researchers using the appropriate functions scored according to the Likert scale and collected open questions to evaluate the comprehensive feeling of ease of use during treatment.
CTCAE level 1 and 2 toxic reaction ratio, Adverse Events (AE) rate, Serious Adverse Events (SAE) rate | screening, 1 months ± 7 days, 2 months ± 7 days, 3 months ± 7 days after the last treatment
  The proportion of subjects who had toxic reactions of levels 1 and 2 during the clinical trial period.The researchers record AE that appeared during the clinical trial cycle and grade it according to CTCAE 5.0
lab test, Eastern Cooperative Oncology Group (ECOG) grade | screening, 1 months ± 7 days, 2 months ± 7 days, 3 months ± 7 days after the last treatment
  Conduct a laboratory examination and the researchers will judge the clinically significant changes in the reporting laboratory indicators. ECOG physical condition grading assessment, and the researchers judge the report of the results clinical significance of the change.
tumor recurrence rate | screening, 1 months ± 7 days, 2 months ± 7 days, 3 months ± 7 days after the last treatment
  The rate of tumor recurrence is the ratio of the number of subjects who have relapsed to the total number of subjects. The CT or MRI imaging changes of tumors before and after treatment will be evaluated by an imaging review team based on RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Yimin Liu, Professor, Study Director — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Shen Fu, Professor, Study Director — Guangzhou Concord Cancer Center
Locations (1):
- Varian ProBeam 360, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No